CLINICAL TRIAL: NCT01266798
Title: Effects of a Patient Directed Web-portal to Improve Health Literacy Skills
Acronym: PREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University of Oslo (Other); Norwegian Knowledge Centre for the Health Services (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REK S-07414b [1.2007.2076]
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Health Behavior
Keywords: Health literacy, participation
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Portal arm (Experimental)
  Interventions: Behavioral: Portal
- Treatment as usal (No Intervention)

INTERVENTIONS:
Behavioral: Portal — The portal was tailored to improve the lay public's' "healthy skepticism", or in other words, critical and social literacy skills to assist patients in the decision-making process and for improving access to health information and participation. Illustrated by typical examples which can be found in the news and through patient stories, the portal provides an introduction to research methods, the underlying principles of science and critical assessment tools appropriate for a lay public.
  1. A checklist for critical assessment of health information
  2. Access to research databases for health information and an introduction to research methods and principles of science
  3. A checklist to the consultation
  Arms: Portal arm

SUMMARY:
Access to the best available evidence, and the ability to obtain and understand such information is seen as necessary to protect the public's interests and critical to empowerment, but is also a precondition for participation in the decision making.

A web portal serving as a generic (non disease- specific) tailored tool was developed in the conceptual framework of shared decision making and evidence based practice to improve the lay- public's critical and social literacy skills and activation. A randomized controlled parallel trial using a simple randomization procedure will be conducted, including 200 parents of children <4 with internet access. Parents will be allocated to receive either the portal or no intervention. Primary and secondary outcomes include: the ability to find research based information, critical appraisal skills, perceived behavioural control, attitudes and perceived pressure associated with searching for information, and participation.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children age <4 will be recruited with access to internet.

Exclusion Criteria:

* Participants will be excluded if one other in the household already participates in the study (due to spill-over effect) and if they do not have children <4.
* Since the recruitment will be done online, there is no need to screen for access to internet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Changes in predictors of search and use of health information | Week 3
  Based on the theory of planned behavioral manual a questionnaire has been developed and validated in order to explore what predictors (efficacy, attitudes and perceived pressure) to search and use of health infomration.

SECONDARY OUTCOMES:
The ability to find reliable answers to a health question | Week 1
  Participants will be asked to formulate a (health) question and to find information that can answer this question. The participants will be asked to copy and paste the internet link to the information they found.The outcome will be evaluated pragmatically by categorizing the information as based on: 1. research or 2. expert advice/ other. The information will be categorized blindly by two independent researchers. The direction of effect is expected to be positive, in that more participants will find research based information than those in the control group.
Critical appraisal of health information | Week 2
  Participants will be asked to rate a piece of health information about childhood vaccination using DISCERNs item number 16. DISCERN is an instrument designed to judge the quality of written information about treatment choices. The mean value rating of the information will be measured against a "standard" rating made by experts on the same information. The direction of effect is predicted to be positive, in that the mean overall score of the intervention group will be closer to the standard than the control group.
Participation (activation) | Week 3
  The patient activation measure (PAM) has been developed to measure activation. The instrument includes 4 domains; believing the patient role is important, having confidence and knowledge necessary to taking action, actually taking action to improve one's health, and staying the course under stress.
Satisfaction with portal | Week 3
  We will also ask participants to comment on satisfaction with the portal after the other data collection has been submitted. This will be done based on the Honeycomb criteria which were also used in the qualitative evaluation. The honeycomb model is a well-renowned and much used instrument to measure user experience

CONTACTS AND LOCATIONS:
Overall Officials: Sølvi Helseth, Professor, Study Director — Oslo University College; Arild Bjørndal, Professor, Study Director — Oslo university; Astrid Austvoll-Dahlgren, MA, Principal Investigator — Oslo University College
Locations (1):
- Oslo University College, Faculty of Nursing, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Austvoll-Dahlgren A, Bjorndal A, Odgaard-Jensen J, Helseth S. Evaluation of a web portal for improving public access to evidence-based health information and health literacy skills: a pragmatic trial. PLoS One. 2012;7(5):e37715. doi: 10.1371/journal.pone.0037715. Epub 2012 May 31. PMID 22701531